CLINICAL TRIAL: NCT03802175
Title: The Application Of Lung Ultrasound About Pulmonary Complications In Postoperative Hypoxemia Patients After General Anesthesia：A Prospective Observational Study
Brief Title: The Application Of Lung Ultrasound In Postoperative Hypoxemia Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-177
Record Dates: First submitted 2019-01-02; First posted 2019-01-14 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-01

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative hypoxemia was persistent and common after surgery.Rapid diagnosis and subsequent therapeutic measures must be adopted by anesthesiologists.Lung ultrasound has been confirmed to be more sensitive and accurate for diagnosis of pulmonary ailment than chest radiography.The primary objective of the present study was to evaluate lung complications by bedside lung ultrasonography on patients suffered from hypoxemia after general anesthesia in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

- at least 18 years of age, hypoxemia after general anesthesia ( definded as a SPO2 <92%,greater than 30s)

Exclusion Criteria:

* Covered with surgical dressings from opening thoracic and breast surgery, noncooperate from schizophrenia or delirium, a BMI higher than 40 kg/m2, unstable hemodynamics, dyspnea from residual opioids or muscle relaxants, hemoglobin of 8g/L or less, risk of bleeding, body temperature was more than 38℃ or less than 36℃

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parients in postoperative care unit(PACU) of 18 years at least and suffering from hypoxemia after general anesthesia and noncardiac surgeries were included in our study.
Sampling Method: Probability Sample
Enrollment: 113 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Complications of Lung Ultrasound | 20 minutes after tracheal extubation
  Pulmonary disease including atelectasis, pneumonia, pneumothorax and pleural effusion would be discovered by lung ultrasound

SECONDARY OUTCOMES:
Comparison of Lung Ultrasound and Computed Tomography(CT) | Within 1 hour after examnation of Lung Ultrasound
  Lung ultrasound offers high sensitivity and specificity when compared with CT

OTHER OUTCOMES:
Correlative Factors of Lung Ultrasound Score | Through study completion, up to 8 months
  Higher score value represent more ventilation loss

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Study Chair — Zhejiang University
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xie C, Sun K, You Y, Ming Y, Yu X, Yu L, Huang J, Yan M. Feasibility and efficacy of lung ultrasound to investigate pulmonary complications in patients who developed postoperative Hypoxaemia-a prospective study. BMC Anesthesiol. 2020 Sep 1;20(1):220. doi: 10.1186/s12871-020-01123-6. PMID 32873237